CLINICAL TRIAL: NCT00486187
Title: Effects of ROSIglitazone on Inflammatory Markers and Adipokines in Diabetic Patients Using an Angiotensin Receptor Blocker (TELmisartan) - The ROSITEL Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Milan Gupta (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Dr. Milan Gupta, MD, Canadian Collaborative Research Network
Organization: Canadian Collaborative Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVD105195
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Thiazolidinediones; Rosiglitazone; Adipokine; Inflammation; Cardiometabolic risk; Angiotensin receptor blocker
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation | interventions — Rosiglitazone; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatment-naive subjects randomly assigned to rosiglitazone (4 mg/day force titrated to 8 mg/day).
  Subjects taking metformin before randomization were randomly assigned to the addition of rosiglitazone (4 mg/day force titrated to 8 mg/day).
  Subjects taking glyburide before randomization were randomly assigned to the addition of rosiglitazone (4 mg/day).
  Interventions: Drug: rosiglitazone
- 2 (Active Comparator): Treatment-naive subjects randomly assigned to metformin (250 mg twice per day [BID] titrated to 500 mg BID if baseline A1C ≥7.5% and ≤8.0%, or 500 mg BID titrated to 1 g BID if baseline A1C >8.0%).
  Subjects taking metformin before randomization were randomly assigned to the addition of glyburide (2.5 mg BID titrated to 5 mg BID if baseline A1C ≥7.5% and ≤8.0%, or 5 mg BID titrated to 10 mg BID if baseline A1C >8.0%).
  Subjects taking glyburide before randomization were randomly assigned to the addition of metformin (250 mg BID titrated to 500 mg BID if baseline A1C ≥7.5% and ≤8.0% or 500 mg BID titrated to 1 g BID if baseline A1C >8.0%).
  Interventions: Drug: metformin or sulfonylurea

INTERVENTIONS:
Drug: rosiglitazone
  Other Names: Avandia
  Arms: 1
Drug: metformin or sulfonylurea
  Arms: 2

SUMMARY:
The purpose of the ROSITEL study is to assess the effects of rosiglitazone, as compared to standard oral therapies for diabetes (metformin/sulfonylurea), on inflammatory markers and adipokine levels in diabetic patients using an angiotensin receptor blocker (ARB).

We hypothesize that ARB-treated diabetic patients receiving rosiglitazone will experience greater reductions in vascular inflammation and levels of leptin and resistin, associated with increased adiponectin levels, compared to a metformin/sulfonylurea regimen, and that these benefits will result in part, from greater improvements in insulin sensitivity in the rosiglitazone group.

DETAILED DESCRIPTION:
Type 2 diabetes is a chronic and progressive disease that is strongly associated with all-cause and cardiovascular mortality. The United Kingdom Prospective Diabetes Study (UKPDS) demonstrated that glycemic control alone only modestly reduces the risk of macrovascular disease among type 2 diabetic patients . Insulin resistance, which has been identified as an important underlying or associated factor in the pathogenesis of type 2 diabetes, is the main proposed mechanism responsible for the accelerated atherosclerosis noted in this population.

Evidence continues to accumulate supporting the role of chronic subclinical vascular inflammation as a central component in the development of atherosclerosis, insulin resistance and type 2 diabetes. Markers of subclinical inflammation, in particular C-reactive protein (CRP) and interleukin-6 (IL-6), have been shown to be independent predictors of both diabetes and cardiovascular risk. More recently, the visceral adipocyte has been recognized to produce a number of metabolically and hormonally active substances, collectively called adipokines. The adipokine adiponectin may have antiatherogenic and anti-inflammatory properties. High levels of adiponectin seem to be associated with protection against type 2 diabetes and atherosclerosis via anti-inflammatory pathways. Unlike adiponectin, leptin and resistin are examples of adipokines that seem to be associated with the development of both atherosclerosis and insulin resistance.

Rosiglitazone is a thiazolidinedione drug that is approved for the treatment of type 2 diabetes. As a nuclear peroxisome proliferator-activated receptor-γ agonist, rosiglitazone reduces insulin resistance, thereby sensitizing the liver, muscle, and adipose tissue to the actions of circulating insulin. Treatment with rosiglitazone has been demonstrated to favourably modify levels of inflammatory biomarkers and adipokines, to attenuate endothelial dysfunction, and to reduce coronary events following percutaneous coronary intervention.

Diabetes and hypertension co-exist in approximately 75% of patients and this combination synergistically augments cardiovascular risk. In fact, blood pressure control seems to be of greater importance in the prevention of macrovascular disease than is glycemic control. Therefore, in patients with diabetes, dual targeting of insulin resistance and blood pressure is essential to reduce overall atherosclerotic risk. Recent evidence suggests that angiotensin receptor blockers (ARB) in addition to their antihypertensive efficacy may directly improve insulin sensitivity. These unique attributes of ARB's may prove particularly beneficial when combined with an insulin sensitizer, such as rosiglitazone, in the treatment of diabetic patients.

The rationale therefore of the ROSITEL study is to compare the effects of rosiglitazone to usual therapy on adipokine levels, inflammatory markers, and insulin sensitivity in ARB-treated diabetic patients with suboptimal glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Hemoglobin A1c (HbA1c) level greater or equal to 0.075
* Treatment naïve (no current oral anti-diabetic therapy) or on monotherapy with either metformin or any sulfonylurea
* Must meet one of the following:

  * Already on an angiotensin receptor blocker (ARB for hypertension and/or microalbuminuria OR
  * If not on an ARB: SBP>129 mm Hg and/or DBP >79 mm Hg And/Or albumin to creatinine ratio (ACR) > 2.0 mg/mmol in men or > 2.8 mg/mmol in women

Exclusion Criteria:

* Women who are pregnant, breast feeding, or not using a reliable method of contraception
* Clinical signs of congestive heart failure or measured left ventricular ejection fraction <40%
* Hemodynamically significant valvular heart disease or hypertrophic obstructive cardiomyopathy
* Insulin-dependent diabetes mellitus
* Use of any PPAR-ỵ agonist (Rosiglitazone or Pioglitazone)
* Renal dysfunction (creatinine > 1.8 x ULN)
* Hepatic disease (liver function test >1.5 x ULN [upper limit normal])
* Other significant laboratory abnormalities that the investigator feels may compromise the patient's safety by participation in the study
* History of systemic inflammatory disease (rheumatoid arthritis, inflammatory bowel disease, systemic lupus erythematous), myositis/myopathic process, or cancer)
* HIV
* Use of steroids or chemotherapy drugs within the past year or chronic use of nonsteroidal anti-inflammatory drugs besides aspirin (use for > 2 weeks within the past year);
* Patients on potassium sparing-diuretics
* Treatment with excluded medications prior to or at the time of randomization
* Known hypersensitivity to Rosiglitazone, or ARB's
* Participation in another clinical study concurrently or within the 30-day phase prior to screening for entry into the present study
* Unwilling to provide written informed consent for study participant and/or
* Unreliability as a study participant as based on the investigator's prior knowledge of the patient, such as the inability or willingness to participate in or complete the study or the presence of concurrent physical or psychological disorders that may make it impractical for the patient to participate in or complete the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change in adiponectin level in the rosiglitazone vs. metformin/sulfonylurea arms | 12 weeks

SECONDARY OUTCOMES:
Secondary end-points include changes in leptin, resistin, hs-CRP, IL-6, MMP-9, ICAM-1, insulin sensitivity (as estimated by the HOMA technique), HbA1c, and lipid levels in the rosiglitazone vs. metformin/sulfonylurea arms | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Milan K Gupta, MD, Principal Investigator — Partners Research
Locations (1):
- Partners Research, Brampton, Ontario, Canada

REFERENCES:
- [Background] Gupta M, Teoh H, Kajil M, Tsigoulis M, Quan A, Braga MF, Verma S. The effects of rosiglitazone on inflammatory biomarkers and adipokines in diabetic, hypertensive patients. Exp Clin Cardiol. 2012 Winter;17(4):191-6. PMID 23592934